CLINICAL TRIAL: NCT03077802
Title: Comparison of Two Needle Insertion Techniques on Success Rate and Complications During Ultrasound Guided Central Venous Catheterization: Seldinger vs. Modified Seldinger Technique
Brief Title: Ultrasound Guided Central Venous Catheterization: Seldinger vs. Modified Seldinger Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1506-126-684
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Catheterization, Central Venous
Keywords: Seldinger technique; Modified Seldinger technique; Complication; Success rate

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Modified Seldinger technique, Experienced group (Experimental): Under ultrasound-guide, we will use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel. The procedure will be performed by experienced practitioner who were defined as board-certified anesthesiologist staffs and had experience of more than 50 central venous catheterizations in both techniques.
  Interventions: Other: Modified Seldinger technique, Experienced group; Other: Long-axis technique; Other: Short-axis technique
- Seldinger technique, Experienced group (Active Comparator): Under ultrasound-guide, the desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. The procedure will be performed by experienced practitioner who were defined as board-certified anesthesiologist staffs and had experience of more than 50 central venous catheterizations in both techniques.
  Interventions: Other: Seldinger technique, Experienced group; Other: Long-axis technique; Other: Short-axis technique
- Modified Seldinger technique, Inexperienced group (Experimental): Under ultrasound-guide, we will use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel. The procedure will be performed by inexperienced practitioner who were junior residents and had experience of less than 50 central venous catheterizations in both techniques.
  Interventions: Other: Modified Seldinger technique, Inexperienced group; Other: Long-axis technique; Other: Short-axis technique
- Seldinger technique, Inexperienced group (Active Comparator): Under ultrasound-guide, the desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. The procedure will be performed by inexperienced practitioner who were junior residents and had experience of less than 50 central venous catheterizations in both techniques.
  Interventions: Other: Seldinger technique, Inexperienced group; Other: Long-axis technique; Other: Short-axis technique

INTERVENTIONS:
Other: Modified Seldinger technique, Experienced group — This is a technique for central venous catheterization. We will use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel. The procedure will be performed by experienced practitioners who are board-certified anesthesiologist staffs and have experience of more than 50 central venous catheterizations in both techniques.
  Arms: Modified Seldinger technique, Experienced group
Other: Seldinger technique, Experienced group — This is a technique for central venous catheterization. The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. The procedure will be performed by experienced practitioners who are board-certified anesthesiologist staffs and have experience of more than 50 central venous catheterizations in both techniques.
  Arms: Seldinger technique, Experienced group
Other: Modified Seldinger technique, Inexperienced group — This is a technique for central venous catheterization. We will use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel. This technique will be performed by inexperienced practitioners who are junior residents and have experience of less than 50 central venous catheterizations in both techniques.
  Arms: Modified Seldinger technique, Inexperienced group
Other: Seldinger technique, Inexperienced group — This is a technique for central venous catheterization. The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. This technique will be performed by inexperienced practitioners who are junior residents and have experience of less than 50 central venous catheterizations in both techniques.
  Arms: Seldinger technique, Inexperienced group
Other: Long-axis technique — Ultrasound probe is placed parallel to the vessel trajectories and needle is advanced using in-plane approach.
Other: Short-axis technique — Ultrasound probe is placed vertical to the vessel trajectories and needle is advanced using out-of-plane approach.

SUMMARY:
The investigators intend to compare the Seldinger technique and modified Seldinger technique on success rate and complications during central venous catheterization by a prospective, randomized, controlled study. The investigators are planning to compare both techniques in both experienced (anesthesiologist board member) and non-experienced practitioners (first and second-grade resident).

DETAILED DESCRIPTION:
Unintended arterial puncture and local hematoma formation are the most common complications during internal jugular vein central venous catheterization. Other serious complications like pseudoaneurysm, arteriovenous fistula, arterial dissection, thrombosis, embolism are also possible. These complications mostly occur by mechanical trauma or injury when advancing needle back and forth to puncture internal jugular vein. Placement of guidewire or dilator can also cause mechanical trauma or injury around the vessel.

Because internal jugular vein collapses easily during needle advance, anterior and posterior wall of the vessel can be punctured simultaneously. Posterior wall puncture can increase the risk of complications of the catheterization. Delicate puncture of the vessel and stable fixation of the needle after puncture are important to reduce overall number of catheterization attempts, increase success rate, reduce complications.

Seldinger technique(thin-wall needle technique) is commonly used procedure to obtain safe access to central vein. The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. Contrarily, modified Seldinger technique(guiding sheath-over-the-needle technique) use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel.

When using Seldinger technique, it is important to fix the needle firmly with hand until the guidewire is placed into the vessel lumen. If hand fixation is not stable, needle tip can migrate from the lumen, can pierce the vessel wall, and carotid artery puncture, and local hematoma formation might occur. Even if there is no evidence of complications, when blood regurgitation fails, overall number of vessel puncture attempts would increase and it is expected that rate of complications of the catheterization would increase.

When using modified Seldinger technique, guiding sheath is easily slid over the needle, providing stable route into the vessel lumen relatively in early step of the catheterization. Therefore, it is expected that stability of the fixation improves, success rate of the catheterization increase, and complications of the catheterization decrease. But there is no high level of evidence yet, and still decision to use which technique is based on experience of the operator.

The investigators are going to compare the Seldinger technique and modified Seldinger technique on success rate and complications during central venous catheterization by prospective, randomized, controlled study.

In addition, any difference in success rate and complications between the two techniques may be different depending on the experience of the practitioners. Therefore, the investigators also plan to compare the two techniques between experienced and non-experienced practitioners.

The success rate and complications between the two techniques may also be different depending on the long and short-axis techniques. As subgroup analyses, we intend to investigate whether there is a difference between Seldinger and modified Seldinger technique according to the experience of the operator or long or short axis approach.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for surgery and internal jugular vein central catheterization

Exclusion Criteria:

* Patient who doesn't agree to the study
* Catheterization site inflammation
* Contralateral diaphragmatic dysfunction
* Anatomic anomalies of carotid artery or vein
* Previous neck surgical history
* Recent (less than 1 month) right internal jugular vein central catheterization

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
number of attempts of needle advance for successful venous puncture | 5 min after internal jugular vein catheterization
  number of attempts of needle advance (number of needling attempt)

SECONDARY OUTCOMES:
incidence of arterial puncture | 5 min after internal jugular vein catheterization
  incidence of arterial puncture during internal jugular vein catheterization
incidence of local hematoma | 5 min after internal jugular vein catheterization
  incidence of jugular venous hematoma during internal jugular vein catheterization
incidence of pneumothorax | 5 min after internal jugular vein catheterization
  incidence of pneumothorax during internal jugular vein
incidence of hemothorax | 5 min after internal jugular vein catheterization
  incidence of hemothorax during internal jugular vein
Time to successful jugular venous catheterization | 5 min after internal jugular vein catheterization
  incidence of hemothorax during internal jugular vein (overall procedure time)
number of attempts of needle advance | 5 min after internal jugular vein catheterization
  number of attempts of needle advance
number of attempts of catheter advance | 5 min after internal jugular vein catheterization
  number of attempts of needle advance (only in modified Seldinger group)
incidence of successful central venous catheterization | 5 min after internal jugular vein catheterization
  incidence of successful central venous catheterization (success defined as completion of catheterization within three attempts of needle advance)
grade of resistance during dilator insertion | 5 min after internal jugular vein catheterization
  grade of resistance during dilator insertion (grade 1: easy, grade 2: moderate, grade 3: difficult, use of blade for skin incision
number of attempts of guidewire advance | 5 min after internal jugular vein catheterization
  number of attempts of guidewire advance through the lumen of needle or guidewire sheath after desired vessel is punctured

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon HK, Hur M, Cho H, Jeong YH, Lee HJ, Yang SM, Kim WH. Effects of practitioner's experience on the clinical performance of ultrasound-guided central venous catheterization: a randomized trial. Sci Rep. 2021 Mar 24;11(1):6726. doi: 10.1038/s41598-021-86322-y. PMID 33762662